CLINICAL TRIAL: NCT05686473
Title: Evaluation of a Treatment Program Based on Psychoeducation of Parents of Children and Adolescents With Fetal Alcohol Spectrum Disorder (FASD)
Brief Title: Psychoeducation of Parents to Children With FASD
Acronym: NorFASDPEdu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NorFASDstudy1
Record Dates: First submitted 2023-01-02; First posted 2023-01-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Fetal Alcohol Spectrum Disorders; Behavior Problem; Adaptive Behavior; Learning Disorders
Keywords: FASD; Psychoeducation; Parenting; Information program
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Mental Disorders; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Assessments with the evaluation measures will be performed at referral to Regional competence centre/inclusion to study (baseline), at admission to the centre 4-5 months later (pre-intervention), and 4-5 months after finishing program (post-intervention). The period between baseline and pre-intervention will be regarded as a control period, in contrast to the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient group (Experimental): Single arm study. The family with child with FASD will act as its own control in the period before intervention starts.
  Interventions: Behavioral: Program of psychoeducation of parents and professionals

INTERVENTIONS:
Behavioral: Program of psychoeducation of parents and professionals — The program consists of a standardized manual-based treatment package as an easily accessible treatment tool for use by professionals in the specialist health services, who have treatment responsibilities for children diagnosed with FASD in Norway.
  The intervention program will last for about 2 months and includes eight sessions, including six digitally based, interactive psychoeducational sessions.
  Topics will be:
  1. General information about FASD
  2. Intervention strategies in kindergartens/schools for children with FASD
  3. Families living with FASD - activities of daily living
  4. Self-regulatory deficits - how to cope
  5. Executive functions in daily life
  6. Social development in children with FASD
  7. Guidance in social settings
  8. Challenging behavior - what can be done

SUMMARY:
By longitudinal, prospective research in children and adolescents with Fetal Alcohol Spectrum Disorders (FASD) and their parents to explore the beneficial effects of participating in a standardized intervention program in order to treat and reduce the consequences of early brain damage. By using elements from international programs based on psychoeducation and parent training, the investigators aim to help parents to better understand and respond to the neurodevelopmental disabilities of their children, and thereby improving behavioral problems and self-regulation deficits.

DETAILED DESCRIPTION:
The main aim of this research project is to evaluate the effects of a standardized intervention program for parents and professionals working with children and adolescents with FASD. Focus will be on care-persons' knowledge and skills and psychoeducation with regard to improved handling of behavioral problems and deficits in self-regulation due to FASD.

To achieve this aim objectives will be:

* to collect and analyse data on family empowerment, parenting skills and stress before and after participation in the intervention program.
* to collect and analyse data on the child's behavior and deficits in self-regulation before and after participation in the intervention program.
* to collect and analyse data on professionals' knowledge of FASD before and after participation in the intervention program.

The current study hypothesizes that caregivers who understand and view their children's behavior from a neurodevelopmental perspective are more likely to feel competence, use antecedent strategies, and thereby reduce child problem behavior and improve functional outcome (Fig. 2). The investigators hypothesize that participation in this program will improve parental empowerment and child self-regulation and behavior compared with baseline assessments.

ELIGIBILITY:
All children and adolescents (age 2,5-18 years) referred to the Regional Competence Centre for children with prenatal alcohol exposure in Arendal, Norway will be invited to participate in the current research project.

Inclusion criteria:

* Valid information about alcohol exposure in fetal life. Exceptions to this inclusion criterion are children who have been adopted and with dysmorphic features that are consistent with full Fetal Alcohol Syndrome.

Exclusion Criteria:

* Children with known genetic syndromes, progressive brain and neuromuscular diseases or major sensory defects (blindness or deafness).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The Children's Global Assessment Scale (CGAS) | up to 10 months
  To evaluate effects of the intervention program well-known standardized, validated measures will be used. Primary outcome measure for the child will be The Children's Global Assessment Scale, which is a numeric scale used by mental health clinicians to rate the general functioning of youths under the age of 18. The scale targets the number of behavioral problems and the frequency of their occurrence.The child or young person is given a single score between 1 and 100. Higher score means better functioning.
The Family Empowerment Scale (FES) | up to 10 months
  Primary outcome measure for parents will be The Family Empowerment Scale to evaluate the magnitude of empowerment in the parent-child system. FES is a 34-item rating scale where the participants rate each item on a 5-point Likert-type rating scale. Scores will range between 34 and 170 points. Increasing scores indicate a positive significance regarding family empowerment.

SECONDARY OUTCOMES:
The Eyberg Child Behavior Inventory (ECBI) | up to 10 months
  In addition, several well-known secondary measures will be used to evaluate additional effects of program. The ECBI questionnaire will be used to evaluate the number of behavioral problems and the frequency of their occurrence before and after the intervention program. ECBI provides a list of 36 problem behaviors commonly reported by parents. The inventory assesses behavior on two dimensions: 1) the frequency of the behavior; 2) whether parents consider it a problem. The frequency ratings range from 1 (never) to 7 (always), and are summed up to arrive at an overall problem behavior Intensity Score, ranging from 36 to 252. Higher score means more behavioral problems.
The Social Responsiveness Scale, Second Edition (SRS-2) | up to 10 months
  The SRS-2 questionnaire will be used to evaluate the severity of social impairment and lack of flexibility in children and adolescents before and after participation in the intervention program. Each domain's T-scores are organized by gender and respondent age, with each domain having varied but similar ranges of possible scores from 32 points-114 points. All T-scores have a mean of 50 points with a standard deviation of 10 points. Higher score means more deficits in social interaction.
The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | up to 10 months
  The BRIEF-2 will be used to evaluate any change in executive functions after participation. Norms tables give T-scores, percentiles, and 90% confidence intervals for four developmental age groups, by gender. Three broad indexes are calculated (Behavior Regulation, Emotion Regulation, and Cognitive Regulation). Higher score means worse outcome.
The Parenting Stress Index (PSI) | up to 10 months
  The PSI questionnaire will be used to evaluate parental stress and load before and after participation in the program.The PSI yields a total score, three domain scores, and 15 subscales. Higher raw scores indicate higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jon S Skranes, Dr Med, Principal Investigator — Sørlandet Hospital HF
Locations (1):
- Sørlandet Hospital, Arendal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Homepage for Regional competence center for children with prenatal alcohol/drug exposure — http://sshf.no/avdelinger/somatikk-arendal/barne-og-ungdomsavdelingen/rkmr